CLINICAL TRIAL: NCT06400550
Title: Identification of Metabolic Phenotypes Associated With Melanoma Metastasis
Status: Recruiting | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Jennifer Gill, ASSISTANT PROFESSOR, University of Texas Southwestern Medical Center
Other Study IDs: STU 052018-031
Record Dates: First submitted 2024-05-01; First posted 2024-05-06 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Melanoma (Skin)
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- 13C-glucose infusion: Tumor samples of patients who receive the optional 13C-glucose infusion will be studied using flux analysis and metabolomic profiling.
- No 13C-glucose infusion: Tumor samples of patients who do not receive the optional 13C-glucose infusion will be studied using metabolomic profiling alone.

SUMMARY:
The goal of this study is to observe metabolic features associated with human melanoma tumors.

DETAILED DESCRIPTION:
This is a single center, correlative study designed to assess metabolic features of melanoma tumors in patients. The study will involve the collection of melanoma tissue at the time of surgical biopsy or excision. All samples will be assessed by mass spectrometry for metabolomic analysis. A subset of patients will have received [U-13C]glucose infusions which will be utilized for isotope tracing metabolic analysis. Relevant clinical data (eg survival, metastasis) will be correlated with metabolic findings.

ELIGIBILITY:
Inclusion Criteria:

* Patients with known or probable malignant melanoma lesions requiring surgical biopsy or excision.
* Subjects of all races and ethnic origins over age 18.

Exclusion Criteria:

* Not a surgical candidate
* Poorly controlled diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years of age with a suspected malignant melanoma
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Glucose Utilisation in the TCA cycle | 5 years
  In patients receiving a [U-13C]Glucose infusion, assess glucose utilization in the TCA cycle by melanoma tumors (defined as fractional enrichment of 13C-label in TCA metabolites)

SECONDARY OUTCOMES:
Relapse free survival | 5 years
  Defined as the time from surgery to disease recurrence or melanoma-related death, whichever occurs first
Overall Survival | 5 years
  Measured as the time of surgery until death from any cause
Development of Lymph Node or Distant Metastasis | 5 years
  Defined as yes/no for each type of metastasis

OTHER OUTCOMES:
Tumor Metabolomic and Lipidomic Profiling | 5 years
  Abundance of metabolites and lipid species, quantified by liquid chromatography mass spectrometry

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Gill, MD, PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No